CLINICAL TRIAL: NCT01425450
Title: A Randomised, Double-blind Placebo-controlled Study to Assess the Safety of Four Single Ascending Doses of HF1020 in Healthy Male Subjects
Brief Title: Safety Study of Four Doses of the Study Drug, HF1020 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trident Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TPI-HF1020-01; 2010-023005-34 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HF1020 (Experimental)
  Interventions: Drug: HF1020
- Placebo (Placebo Comparator)
  Interventions: Drug: HF1020 placebo

INTERVENTIONS:
Drug: HF1020 — Single doses at 0.5 mg capsules, 2.5 mg capsules, 10 mg capsules, and 25 mg capsules in each of cohorts 1, 2, 3 and 4 respectively.
  Arms: HF1020
Drug: HF1020 placebo — Single dose: HF1020 placebo capsule
  Arms: Placebo

SUMMARY:
The study aims to:

* study the safety of the drug (HF1020) in healthy male adults
* study how well the study drug (HF1020) is tolerated in healthy male adults
* find the maximum dose that is tolerated in healthy male adults

DETAILED DESCRIPTION:
This is a single-centre, randomised, double-blind, placebo-controlled, ascending dose study.

Male subjects will be randomised to give a total of 32 evaluable subjects.

Subjects will be sequentially enrolled into 4 cohorts of ascending dose.

Subjects in Cohort 1 will be randomised to receive 0.5 milligrams (mg) HF1020 or placebo (ratio 3:1). When at least 8 subjects within the cohort have completed Day 2 procedures (i.e. Day 1 + 24 hours) and all ongoing subjects have completed the final Day 15 visit, a Safety Review Committee (SRC) will meet, review all safety data prior to dose escalation to the next cohort.

Subjects in Cohort 2 will be randomised to receive 2.5 mg HF1020 or placebo.

Subjects in Cohort 3 will be randomised to receive 10mg HF1020 or placebo.

Subjects in Cohort 4 will be randomised to receive 25mg HF1020 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male
* Subject is aged between 18 and 65 years inclusive
* Subject is able and willing to provide signed informed consent
* Subject's body mass index (BMI) is between 18 and 32 kg/m2 inclusive
* Non-smokers or ex smokers (greater than 1 year) with less than a 5 pack/year history
* Subject's medical history is considered normal in the opinion of the Investigator, with no clinically significant abnormalities. No history of asthma and any concurrent clinically significant illness or concomitant medication use (with the exception of paracetamol and Non-Steroidal anti-inflammatory drugs (NSAIDs) taken as needed during the study).
* Subject is considered to be in good health in the opinion of the Investigator. Normal/clinically acceptable vital signs (blood pressure (systolic blood pressure 100-140mmHg, diastolic blood pressure 60-90mmHg; heart rate 40-100bpm), physical examination and Electrocardiogram (ECG), as determined by the Investigator.
* Subject's screening and pre dose clinical laboratory findings are within normal range or if outside the normal range not deemed clinically significant in the opinion of the Investigator. Lymphocyte subsets must be within normal limits
* QTcB should be less than or equal to 450 msec at screening and pre-dose
* Subject must be willing to abstain from alcohol for 48 hours prior to admission to the unit (including screening visits) and until discharge from the CRU.
* Subjects must be willing to abstain from grapefruit, grapefruit-containing products, cranberry juice, Seville oranges, marmalade or pomelos for 7 days prior to screen and for their participation on the study.
* Subjects must be willing to abstain from exercise more strenuous than walking, 48 hours prior to study visits
* Subjects must be willing to avoid sperm donation and to abstain from actively planning pregnancy during and for three months after the end of the study.
* Male subjects with female partners of child bearing potential must use 2 different forms of highly effective contraception throughout the study; established use of oral, injected/implanted hormonal contraception; placement of an intrauterine device or intrauterine system; use of a barrier method of contraception (condom or occlusive cap with use of a spermicide); male sterilisation (post-vasectomy documentation of the absence of sperm in the ejaculate must be provided). Female partners should not be pregnant or breastfeeding. Subjects are required to continue to use the same contraceptive method for 3 months after their final study visit. In addition, all sexually active subjects must use a condom irrespective of sex of partner or child-bearing potential of partner and even if vasectomised, during the study and for three months after final study visit.
* Forced Expiratory Volume in one second (FEV1) and Forced Vital Capacity (FVC) greater than or equal to 80 % of predicted normal value at Screening Visit
* FEV1/FVC ratio greater than or equal to 0.70 at Screening Visit
* Subject must be willing to remain in the Clinical Research Unit (CRU) for a minimum of two nights.
* Subjects must be able to communicate well with the Investigator, to understand and comply with the requirements and restrictions of the study, and understand and sign the written informed consent

Exclusion Criteria:

* Subject has had a clinically significant illness in the four weeks before screening or during the run-in period
* Subject has a significant history of drug/solvent abuse (within two years prior to Day 1), or a positive drugs of abuse test at screening or prior to randomisation
* Subject with a history of alcohol abuse or currently drinks in excess of 28 units per week, or has a positive breath alcohol test at the Screening Visit or prior to randomisation
* Subject is, in the opinion of the Investigator, not suitable to participate in the study
* Subject who has participated in any clinical study with receipt of an investigational drug within 3 months prior to Day 1
* Subject who has a positive result of human immunodeficiency virus (HIV) Hepatitis B or Hepatitis C screen
* Subject has had a serious adverse reaction or significant hypersensitivity to any drug
* Subject has donated 500 ml or more of blood, or experienced blood loss of 500 ml or more, within 3 months prior to Day 1; or has donated plasma within 7 days prior to Day 1
* Any condition that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs
* Considering or scheduled to undergo any surgical procedure during the duration of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to day 15
  All Adverse events occuring from consent until subject completion will be reviewed at each clinic visit. Subjects will be questioned regarding any events that may have occured between clinic vists.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicines Evaluation Unit, Manchester, Lancashire, United Kingdom